CLINICAL TRIAL: NCT06497959
Title: Contribution of Contrast-Enhanced Ultrasound (CES) in the Fetal-placental Circulation Study
Brief Title: Study of Placental Vascularization Using Contrast Ultrasound
Acronym: EVUPACUS
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Central Hospital, Nancy, France (Other)
Responsible Party: Principal Investigator, Matthieu DAP, Doctor in medicine (Gynaecologist-Obstetrician), Central Hospital, Nancy, France
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 2021PI062; 2023-506936-34-00 (EU CTIS Number)
Record Dates: First submitted 2024-06-20; First posted 2024-07-12 (Actual); Last update posted 2025-05-31 (Actual); Status verified 2025-04

CONDITIONS: Fetal Growth Restriction
Keywords: Contrast-Enhanced Ultrasound (CES)
MeSH Terms: conditions — Fetal Growth Retardation | interventions — contrast agent BR1

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Non-growth restriction group (control group) (Experimental): Fetuses not affected by growth pathology, defined by an estimated weight greater than the 10th percentile at ultrasound
  Interventions: Drug: SonoVue
- Severe growth restriction group (Experimental): Severe growth restriction defined by an estimated fetal weight below the 3rd percentile on ultrasound
  Interventions: Drug: SonoVue

INTERVENTIONS:
Drug: SonoVue — Placental contrast ultrasound using SonoVue by maternal intravenous injection

SUMMARY:
Preeclampsia and intrauterine growth restriction (IUGR) are two principal complications of pregnancy. These diseases are related to placental dysfunction nevertheless knowledge of its pathophysiological mechanisms remains inadequate.

No etiological treatment for these pathologies is available. Inducing birth is the only way to prevent the occurrence of these complications (such as fetal death in utero.

Therefore, a better understanding of placental vascularization under pathological and physiological conditions is necessary. This placental vascularization evolves throughout gestation. Histological studies have improved our knowledge of placental vascular pathologies; however, these are ex vivo data that only provide an incomplete reflection of placental function. In vivo placental studies are therefore essential to understand the mechanisms of placental perfusion. Currently, these studies are limited because the available tools (such as placental Doppler) do not allow for the separate study of maternal placental flow from fetal flow. However, histological evidence clearly establishes maternal placental vascular involvement in IUGR. It would therefore be interesting to study maternal and fetal placental vascularization separately. The development of new in vivo imaging exploration techniques will help to better understand placental pathologies.

In obstetrics, CES would offer the opportunity to study in vivo placental vascularization in a segmented manner (maternal versus fetal side independently) since the microbubbles do not cross the placental barrier. Animal studies show no toxic effects on fetal development nor any crossing of the placental barrier. In humans, the innovative use of this contrast agent has allowed for a better understanding of placental vascularization in the first trimester of pregnancy.

DETAILED DESCRIPTION:
The primary objective is to compare placental contrast ultrasound in patients with medical termination of pregnancy at gestational age 16 weeks - 38 weeks+ 6 days between two groups: the fetal growth restriction one and the no fetal growth restriction.

Methods and analysis: This is a monocentric, prospective comparative, non-randomized, feasibility, open and interventional study. The investigators will include 30 women with medical termination of pregnancy divided in two groups: fetal growth restriction one and the no fetal growth restriction. Women are informed and recruited in the Fetal Medicine units in Nancy, over a period of 48 months.

ELIGIBILITY:
Inclusion Criteria:

* Adult woman (age ≥18 years),
* Gestational age between 16 GW + 0 days and 38 GW + 6 days,
* Singleton pregnancy,
* Whose request of a medical termination of pregnancy (IMG) has been formulated and accepted in a written form by the Centre Pluridisciplinaire de Diagnostic Prénatal (CPDPN) of the Centre Hospitalier Régional Universaitaire (CHRU) de Nancy,
* Affiliated to the social security system or benefit from such a system,
* Having received full information and having signed an informed consent form.

Criteria specific to patients in the "growth restriction" group:

- Severe growth restriction defined by an estimation of foetal weight below the 3rd percentile using ultrasound performed no more than 15 days prior to the IMG (the diagnosis must be established at the time of the request for IMG in routine care).

Exclusion Criteria:

* Person who do not speak French
* Any medical condition contraindicating the administration of SonoVue, in particular:

  * Hypersensitivity to sulfur hexafluoride or to one of the other components of SonoVue® such as polyethylene glycol (PEG),
  * Women with recent acute coronary syndrome or unstable ischaemic heart disease,
  * Women with a right-to-left shunt, severe pulmonary arterial hypertension (pulmonary arterial pressure > 90 mmHg), uncontrolled systemic hypertension and women suffering from respiratory distress syndrome.
* Persons covered by articles L. 1121-5, L. 1121-7 and L1121-8 of the French Public Health Code:

  * Breast-feeding mother
  * Minor (not emancipated)
  * An adult subject to a legal protection (guardianship, curatorship, safeguard of justice)
  * An adult unable to give consent
* Persons deprived of their liberty by a judicial or administrative decision, persons under psychiatric care by virtue of articles L. 3212-1 and L. 3213-1

Ages: 18 Years to 64 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 30 (Estimated)
Dates: Start 2025-04-09 (Actual); Primary Completion 2029-04-09 (Estimated); Study Completion 2029-04-10 (Estimated)

PRIMARY OUTCOMES:
The measurement of signal strength | 1 day
  The measurement of signal strength (in arbitrary units) in the Inter-Villi Space of the placetna ,obtained by contrast ultrasound, in women who have confirmed a medical termination of pregnancy according to the group defined by fetal weight in percentile as a function of term. Severe Intrauterine Growth Restriction (IUGR) is defined as a weight below the 3rd percentile for gestational age.For each group, these parameters will be obtained by qualitative analysis (i.e. presence/absence of contrast medium passage) and semi-quantitative analysis (enhancement percentage, area under the curve, time to peak, slopes -wash-in rate and wash-out rate, etc.) using dedicated software VueBox, BRACCO

SECONDARY OUTCOMES:
Measurement of the vascularization parameters of the Inter-Villi Space: infusion kinetics. | 1 day
  Measurement of the vascularization parameters of the Inter-Villi Space : infusion kinetics by ultrasound with a contrast agent: SonoVue ®.
Measurement of the vascularization parameters of the umbilical cord: infusion kinetics | 1 day
  Measurement of the vascularization parameters of the umbilical cord: infusion kinetics by ultrasound with a contrast agent: SonoVue ®.
Measurement of the placenta vascularization using histological analysis | through study completion, on average of 24 months
  Measurement of the placenta vascularization using histological analysis according to the Amsterdam Standardised Analysis criteria.
Comparison of of the placenta vascularization using histological analysis and the measurement of the vascularization parameters of the Inver-Villi Space. | through study completion, on average of 24 months
  Measurement of the placenta vascularization using histological analysis according to the Amsterdam Standardised Analysis criteria and the vascularization parameters of the umbilical cord: infusion kinetics by ultrasound with a contrast agent: SonoVue ®.

CONTACTS AND LOCATIONS:
Locations (1):
- CHRU de NANCY, Nancy, France

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data (IPD) will be made available upon reasonable request, after de-identification.
  Additional documents such as the statistical analysis plan may also be available.
  Data will be available starting 3 months after publication and for a period of 5 years.
  Researchers must submit a methodologically sound proposal reviewed and approved by an independent ethics committee.
  Data will be shared via a secure online platform and under a data access agreement.
  Requests should be addressed to the corresponding author: Dr. Matthieu Dap (m.dap@chru-nancy.fr)

REFERENCES:
- [Derived] Lefebvre J, Cherifi A, Hossu G, Fijean AL, Morel O, Bertholdt C, Beaumont M, Dap M. Contributions of contrast-enhanced ultrasound (CEUS) to a fetal-placental circulation study (EVUPACUS): a protocol for a prospective comparative study in a population of women undergoing termination of pregnancy. BMJ Open. 2025 Aug 10;15(8):e093090. doi: 10.1136/bmjopen-2024-093090. PMID 40784773